CLINICAL TRIAL: NCT06186687
Title: Rehabilitative Approaches: Myofunctional Therapy and Retropalatal Narrowing and Snoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKFR-202312.01
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Snoring; Pharyngeal Collapse
Keywords: Myofunctional therapy exercise; pharyngeal area collapse; snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myofunctional Therapy Exercise (Experimental): Seventeen patients whom already diagnosed by an Ear, Nose and Throat specialist as having risk of obstructive sleep apnea based on the questionnaire and FN study that showed pharyngeal muscle collapse in the pharyngeal area (velopharyngeal area/retropalatal), performed MT two times per day for 20 minutes every day for six weeks. Exercises were performed at home with monitoring by the exercise log book, submitting a clear video of each exercise, and being evaluated once a week by the doctor. Patient compliance was classified as good if the patient performed >75% of the exercises weekly. This study evaluated the velopharynx/retropalatal area (with FN), symptoms of daytime sleepiness with the Epworth Sleepiness Scale (ESS) questionnaire, and snoring intensity and frequency taken from the Berlin questionnaire that were filled out before and after undergoing training for 6 weeks.
  Interventions: Behavioral: Myofunctional therapy exercise

INTERVENTIONS:
Behavioral: Myofunctional therapy exercise — Myofunctional therapy involves various exercises to train muscles in the soft palate, tongue, face, and pharynx. Vocal letters are used to train the palatopharyngeus, palatoglossus, uvula, tensor veli palatine, and levator veli palatine muscles. Tongue exercises involve sliding the tongue to the upper and side surfaces of the teeth, placing the tip in front of the palate, and pressing and sucking the tongue up to the palate. Face exercises involve inflating the cheeks, gargling, and sucking the cheeks to exercise the orbicularis oris muscle and the buccinator muscle. Icing stimulates the mouth, producing a cold, chilling, and numbing effect, causing reflexive contraction of the palate, tongue, and pharyngeal muscles.

SUMMARY:
Sleep is an important activity and snoring is the most often reported complaint. Snoring is also very common in the general population. Moreover, snoring can negatively impact bed companions' quality of sleep, daytime sleepiness, strain of relationships, social embarrassment and disturb mental health that in the end will reduce quality of life. Anatomical risk factors are believed to be one of major contributors to upper airway constriction during sleep. Treatment for this condition include lifestyle modifications (such as quitting alcohol or losing weight), positional therapy, mandibular advancement devices, upper airway surgery, and nasal continuous positive airway pressure. Myofunctional therapy (MT) as an adjunctive or alternative therapy can lower Apnea-Hypopnea Index in obstructive sleep apnea patients with pharyngeal dilator muscle collapse. Although these may be beneficial, the impact of MT on retropalatal narrowing as one of the snoring causes needs to be better established. This study was done to find out the impact of MT in people with snoring who have a collapsed pharynx that is located by a Flexible nasolaryngoscopy.

DETAILED DESCRIPTION:
Sleep is an important activity; it makes up one-third of a person's life, and in sleep medicine clinics, snoring is the most often reported complaint. Snoring is also very common in the general population. Studies indicate that women have a higher incidence of this condition above 65 years, increasing after menopause, while men experience it between 45 and 64 years of age. While snoring may be a predictor of the more serious condition of obstructive sleep apnea, primary snoring is common. Moreover, snoring can negatively impact bed companions' quality of sleep, daytime sleepiness, strain of relationships, social embarrassment and disturb mental health that in the end will reduce quality of life. Anatomical risk factors are believed to be one of major contributors to upper airway constriction during sleep. Pharyngeal narrowing can be facilitated by anatomic characteristics such as a large neck circumference, soft tissue, bone, or arteries. Flexible nasolaryngoscopy (FN) is an alternative diagnosis to direct viewing of the airway, from the nasal cavity to the larynx area. Aside from being easier to perform and more affordable, a complete examination of the airway can identify the location of the pharyngeal narrowing that causes obstruction more specifically. Treatment for this condition include lifestyle modifications (such as quitting alcohol or losing weight), positional therapy, mandibular advancement devices, upper airway surgery, and nasal continuous positive airway pressure are among the treatments for treating snoring. Myofunctional therapy (MT) as an adjunctive or alternative therapy can lower Apnea-Hypopnea Index in obstructive sleep apnea patients with pharyngeal dilator muscle collapse. The exercises are non-invasive, cost-effective, and have physiological characteristics. Improvement in upper airway obstruction is supported by improvements in upper airway muscle tone. Although these may be beneficial, the impact of MT on retropalatal narrowing as one of the snoring causes needs to be better established. This study was done to find out the impact of MT in people with snoring who have a collapsed pharynx that is located by a FN.

ELIGIBILITY:
Inclusion Criteria:

* high risk of OSA (STOP-Bang questionnaire ≥ 3 and Berlin Questionnaire score positive in ≥ 2 category)
* Already diagnosed by an Ear, Nose and Throat specialist as having risk of obstructive sleep apnea based on the questionnaire and FN study that showed pharyngeal muscle collapse in the pharyngeal area (velopharyngeal area/retropalatal)

Exclusion Criteria:

* history of lung disease,
* craniofacial anatomy abnormalities,
* consuming drugs with sedative effects, alcohol, anti-depressants, or anti-anxiety groups in the last 3 months before

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Widening of retropalatal area | 6 weeks
  The retropalatal area was evaluated with flexible nasolaryngoscopy before and after 6 weeks of myofunctional therapy exercise.
Symptoms of daytime sleepiness | 6 weeks
  Symptoms of daytime sleepiness was evaluated with Epworth Sleepiness Scale (ESS) score before and after 6 weeks of myofunctional therapy exercise. The minimum values of the socre is 0 and the maximum value is 24. The higher the ESS score, the higher their 'daytime sleepiness', which gives a worse outcome.
Snoring intensity and frequency | 6 weeks
  Snoring intensity and frequency evaluation were taken from the Berlin questionnaire before and after 6 weeks of myofunctional therapy exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Vitriana Biben, Dr; MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia